CLINICAL TRIAL: NCT02887638
Title: Posture-related Headache: Profile Analysis and Intervention
Brief Title: Headache Analysis and Intervention
Acronym: PRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other); Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other); Orbisch Medisch Centrum (Unknown); Zuyd University of Applied Sciences (Other); Algemeen Ziekenhuis Vesalius (Other)
Responsible Party: Principal Investigator, prof. dr. Marita Granitzer, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHA-2016
Record Dates: First submitted 2016-08-19; First posted 2016-09-02 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Headache
Keywords: posture, sit
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- headache (Experimental): Patients diagnosed (neurologist - anesthesiologist - manual therapist) with tension-type and/or cervicogenic headache. During a first phase the sitting-posture, dura mater profile and pain-profile of the Headache-group will be analyzed. In a second phase, the patients will be sub-classified according to the data-analysis and receive intervention (Individual Profile Analysis +Physical therapy Intervention)
  Interventions: Other: Individual Profile Analysis (Physical therapy Intervention)
- asymptomatic controls (No Intervention): Asymptomatic controls, matched for gender and age. During a first phase the sitting-posture, dura mater profile and pain-profile of the control-group will be analyzed.

INTERVENTIONS:
Other: Individual Profile Analysis (Physical therapy Intervention) — The Individual Profile Analysis consists of the following components:
  * Analysis of the sitting-posture profile:
    o cervical spine, thoracic spine, lumbar spine and pelvis during a longitudinal provoking task (working at a laptop).
  * Analysis of the dural profile before and after the provoking task:
    o Determination of the dural sensitivity by the use of the slump-test
  * Analysis of the pain profile before and after the provoking task:
    * Determination of pressure pain sensitivity by the use of pressure algometry
    * Determination of the influence of pain on the quality of life by the use of the HIT-6 questionnaire
  Arms: headache

SUMMARY:
Diagnosing and treating posture-related headache (PRH), such as tension-type and cervicogenic headache, is seriously hampered because of common features and complex interaction of the neurological and musculoskeletal system. Current therapies are therefore not as effective and the population of patients with PRH keeps on increasing. The diagnostic as well as the therapeutic process need more structure in order to select the most effective treatment; thereby contributing to preventive measures. This goal can be achieved through fundamental research with a clinically oriented background. Our study starts from a clinical problem, with a growing incidence, and is therefore highly relevant. Because sitting-posture seems to play an important role in PRH, the first step in the diagnostic process is to analyse postural differences between a PRH- and a control-group. In addition, the role of the dura mater in the headache-process will be examined. Patients with PRH will be classified in homogeneous groups based on these results. In a second phase individual-specific treatment programs will be composed. The general treatment-approach of postural abnormalities in the past failed because of the heterogeneous patient-populations. Sub-classifying musculoskeletal problems has been proven to be successful in the past (O'Sullivan & Dankaerts, non-specific low back pain).

Our study is divided in 2 phases:

* phase 1: profile analysis (no intervention, experimental headache-group vs. asymptomatic controls)
* phase 2: interventional phase (clustered headache-groups, based on the results of phase 1

ELIGIBILITY:
Inclusion Criteria Headache-group:

1. Males and females between 20 and 50 years
2. Confirmed medical diagnosis of tension-type headache, cervicogenic headache or a mixture
3. Headache can be provoked by awkward cervical and/or head postures

Exclusion Criteria Headache-group:

1. Pregnancy
2. History of pericranial surgery
3. Serious pathology (neurological/cardiovascular/endocrine/musculoskeletal)
4. Red flags
5. Physical or manual therapy treatment for headache < 4 weeks prior the study
6. Excessive (> 10 days/month for > 3 months) use of: ergotamine, NSAID's, opioids, triptans, acetylsalicylic acid and simple analgesics
7. Psychiatric comorbidity
8. Visual or temporo-mandibular dysfunction

Inclusion Criteria Control-group:

1. Males and females between 20 and 50 years
2. Asymptomatic, no headache-history

Exclusion Criteria Control-group:

1. Pregnancy
2. History of pericranial surgery
3. Excessive (> 10 days/month for > 3 months) use of: ergotamine, NSAID's, opioids, triptans, acetylsalicylic acid and simple analgesics
4. Visual or temporo-mandibular dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Sitting-posture-profile | day 1
  Sitting-posture will be measured with a 3D-video analysis (Bonita, ©Vicon Motion Systems Ltd. UK). Markers are placed on specific anatomical reference points on the participant. Afterwards angles (°) will be automatically calculated (Nexus, ©Vicon Motion Systems Ltd. UK)
Pain-Profile | day 1
  'Pain Pressure Threshold' will be measured. Through pressure- algometry (a) 'Pressure Pain Detection Threshold' (kPa/cm²) and (b) 'Pressure Pain Tolerance' (sec) will be determined (Somedic Sales AB, Stockholm Sweden).
Sitting-posture-profile | week 1 up to week 8
  Sitting-posture will be measured with a 3D-video analysis (Bonita, ©Vicon Motion Systems Ltd. UK). Markers are placed on specific anatomical reference points on the participant. Afterwards angles (°) will be automatically calculated (Nexus, ©Vicon Motion Systems Ltd. UK)

SECONDARY OUTCOMES:
Headache-related medication-use, headache intensity, duration and frequency. | week -4 up to week 8
  Through the use of a specific diary the secondary outcomes will be evaluated.
Impact of headache on the quality of life. | week -4 up to week 8
  The 'Headache Impact Test (HIT-6)' will be used.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (3):
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - Leuven University, Leuven
- Netherlands (2):
  - Zuyd University, Heerlen
  - Orbis Medisch Centrum, Sittard

IPD SHARING:
Plan to Share IPD: Undecided